CLINICAL TRIAL: NCT06128798
Title: A Randomized Controlled Trial on Effect of Preoperative Immunonutrition Versus Standard Oral Nutrition in Patient Undergoing Colorectal Surgery.
Brief Title: Effect of Preoperative Immunonutrition Versus Standard Oral Nutrition in Patient Undergoing Colorectal Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Manivaasan Pannirselvam, Dr Manivaasan Pannirselvam, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: USM/JEPeM/KK/23050402
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Neoplasms
Keywords: Immunonutrition; Colorectal Cancer; Oral Impact
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Impact (Experimental): Immunonutrition enriched with omega-3 fatty acids, arginine, nucleotides, and soluble fibre. Main source of protein is arginine and casein.
  Interventions: Dietary Supplement: Oral Impact
- Nutren Optimum (Active Comparator): A balanced nutritional supplement that enhance body natural defence and support recovery during illness.
  Interventions: Dietary Supplement: Nutren Optimum

INTERVENTIONS:
Dietary Supplement: Oral Impact — A serving of 74 gm (containing 309 kcal ) of oral impact mixed with 250 ml of water. Each participant will receive total of 3 servings daily for 7 days pre operatively .
  Arms: Oral Impact
Dietary Supplement: Nutren Optimum — A serving of 66.8 gm ( containing 304 kcal ) of nutren optimum mixed with 300 ml of water.Each participant will receive total of 3 servings daily for 7 days pre operatively .
  Arms: Nutren Optimum

SUMMARY:
This is a randomised controlled clinical trial . The investigators aim to compare the effects of preoperative immune modulating enteral nutrition and standard oral nutrition supplement on clinical outcomes of the patients undergo colorectal cancer surgery.

The main questions it aims to answer are:

1. Does immunonutrition preoperatively facilitate earlier return of Gastrointestinal function?
2. Does immunonutrition significantly reduce risk of post-operative surgical site infections?
3. Does immunonutrition significantly reduce duration of hospital stay in patients undergoing colorectal surgery?

Immunonutrition can be defined as modulation of either the activity of the immune system, or modulation of the consequences of activation of the immune system, by nutrients or specific food items fed in amounts above those normally encountered in the diet.

Oral IMPACT is readily available immunonutrition consist of 3.3 g of arginine,0.8 g of omega-3 fatty acids and 3.0 g of nucleotides per servings.

Nutren Optimum is a balanced nutritional supplement that enhance body natural defence and support recovery during illness. However, it does not consist all the component of immunonutritons. Hence , Oral IMPACT will be used as study sample on experimental arm whereas Nutren optimum will be used as study sample on control arm.

Partipicant will be randomised into this two arm and then they will consume the respective arm study material for total of 7 days preoperatively.

Data will be collected in post operative period and will be analysed.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the commonest cancer in Malaysian men and the second most common cancer in Malaysian women, accounting for age standardized rate of 14.8 and 11.1 incidences per 100,000 population respectively.

Oncological colonic resection is one of mainstay treatment modality for colorectal tumour. Major surgery precipitate release of stress hormones, inflammatory mediators and metabolic changes resulting in significant catabolic phenomena. This sequentially imposed significant dysfunction of the overall host homeostasis, defence mechanism and inflammatory response. Hence, the major setbacks of colorectal surgery are delay return of normal bowel physiology state, post-operative complications and prolonged hospital stay. This affects patients physiologically and psychologically.

Traditionally , patients undergo major abdominal surgery will be kept nil per oral for 6 to 12 hours prior to operation. Post operatively, parenteral or enteral fluids given until bowel function returns to normal. Fortunately, the introduction of the Enhanced Recovery After Surgery (ERAS) programs in last decade has led to enhanced in the recovery of patients postoperatively. The main aspects of substantial improvements in the care of postoperative patients include early initiation of oral intake as soon as possible, integration of nutrition support ,metabolic control and early mobilisation.

As nutritional status plays a significant role to influence the clinical outcomes, nutrition support has been widely used for elective colorectal surgery patients. Literature reported that nutritional risk rate of cancer patients to be 26% to 76 %, higher than of general patients.

Immunonutrition has been used as therapeutic options for peri-operative nutritional management in patients undergoing surgery. The nutrients of immunonutrition formula usually include arginine, omega-3 fatty acids, glutamine and nucleotides.

The current international guidelines recommend that patient's with high risk of malnutrition should be given immunonutrition in perioperative period prior to major oncologic surgeries.These guidelines are based on randomized controlled trials demonstrating a reduction in the rate of post-operative complications.

Oral IMPACT is readily available immunonutrition consist of 3.3 g of arginine,0.8 g of omega-3 fatty acids and 3.0 g of nucleotides per servings. It comes in sachet form which mixed with water prior to consumption. Multiple randomised controlled trial supported Oral IMPACT as immunonutrition.

Nutren Optimum is a balanced nutritional supplement that enhance body natural defence and support recovery during illness. However, it does not consist all the component of immunonutritons. Hence , Oral IMPACT will be used as study sample on experimental arm whereas Nutren optimum will be used as study sample on control arm.

In nutshell , it is important for proper perioperative nutritional support for patients scheduled for colorectal surgery. It remain as major advantage for successful procedure.

In the light of this guideline investigators aimed to compare the effects of preoperative immune modulating enteral nutrition and standard oral nutrition supplement on clinical outcomes of the patients undergo colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age is at least 18 years old
2. All cases posted for Laparoscopic elective colorectal surgery

Exclusion Criteria:

1. Known allergy to milk, fish, and soy.
2. On fluid restriction
3. Emergency Surgery
4. Minor Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Physiology Return of Bowel Function | Through study completion , an average of 1 year
  To compare the time of the first flatus and first bowel evacuation between Oral Impact® and Nutren Optimum ® when consumed in the preoperative in those undergoing colorectal surgery.

SECONDARY OUTCOMES:
Surgical Site Infection | 30 days post operative period
  To associate the difference on post operative surgical site infection in between those consuming Oral Impact® versus Nutren Optimum ® in the preoperative period after colorectal surgery.
Length of Hospital Stay | From date of admission until patient is discharged back home or date of death from any cause during admission , whichever come first ,accessed up to 1 year
  To study on the differences on duration of hospital stay after colorectal surgery in those consuming Oral Impact® and Nutren Optimum ®

CONTACTS AND LOCATIONS:
Overall Officials: Siti Rahmah Binti Hashim Isa Merican, Dr, Study Director — Hospital Universiti Sains Malaysia; Muhammad Faeid BIn Othman, Dr, Study Director — Hospital Universiti Sains Malaysia; Manivaasan Pannirselvam, Dr, Principal Investigator — Hospital Universiti Sains Malaysia; Nor Syarahani Binti Jusoh, Dr, Study Director — Hospital Universiti Sains Malaysia; Wong Pak Kai ( Michael), Dr, Study Director — Hospital Universiti Sains Malaysia
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months after Publication
Access Criteria: Primary Investigator ; Sub-Investigator

REFERENCES:
- [Background] Shaikh SR, Jolly CA, Chapkin RS. n-3 Polyunsaturated fatty acids exert immunomodulatory effects on lymphocytes by targeting plasma membrane molecular organization. Mol Aspects Med. 2012 Feb;33(1):46-54. doi: 10.1016/j.mam.2011.10.002. Epub 2011 Oct 19. PMID 22020145
- [Result] Fearon KC, Ljungqvist O, Von Meyenfeldt M, Revhaug A, Dejong CH, Lassen K, Nygren J, Hausel J, Soop M, Andersen J, Kehlet H. Enhanced recovery after surgery: a consensus review of clinical care for patients undergoing colonic resection. Clin Nutr. 2005 Jun;24(3):466-77. doi: 10.1016/j.clnu.2005.02.002. Epub 2005 Apr 21. PMID 15896435
- [Result] Lee SY, Jung MR, Kim CH, Kim YJ, Kim HR. Nutritional risk screening score is an independent predictive factor of anastomotic leakage after rectal cancer surgery. Eur J Clin Nutr. 2018 Apr;72(4):489-495. doi: 10.1038/s41430-018-0112-3. Epub 2018 Feb 19. PMID 29459787
- [Result] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Result] Chang HR, Bistrian B. The role of cytokines in the catabolic consequences of infection and injury. JPEN J Parenter Enteral Nutr. 1998 May-Jun;22(3):156-66. doi: 10.1177/0148607198022003156. PMID 9586794
- [Result] Klek S, Szybinski P, Szczepanek K. Perioperative immunonutrition in surgical cancer patients: a summary of a decade of research. World J Surg. 2014 Apr;38(4):803-12. doi: 10.1007/s00268-013-2323-z. PMID 24178185
- [Result] Grimble RF. Basics in clinical nutrition: Immunonutrition - Nutrients which influence immunity: Effect and mechanism of action. Vol. 4, e-SPEN. Elsevier BV; 2009.
- [Result] Xiong L, Teng JL, Botelho MG, Lo RC, Lau SK, Woo PC. Arginine Metabolism in Bacterial Pathogenesis and Cancer Therapy. Int J Mol Sci. 2016 Mar 11;17(3):363. doi: 10.3390/ijms17030363. PMID 26978353
- [Result] Braga M, Gianotti L, Vignali A, Carlo VD. Preoperative oral arginine and n-3 fatty acid supplementation improves the immunometabolic host response and outcome after colorectal resection for cancer. Surgery. 2002 Nov;132(5):805-14. doi: 10.1067/msy.2002.128350. PMID 12464864
- [Result] Hess JR, Greenberg NA. The role of nucleotides in the immune and gastrointestinal systems: potential clinical applications. Nutr Clin Pract. 2012 Apr;27(2):281-94. doi: 10.1177/0884533611434933. Epub 2012 Mar 5. PMID 22392907
- [Result] Novak F, Heyland DK, Avenell A, Drover JW, Su X. Glutamine supplementation in serious illness: a systematic review of the evidence. Crit Care Med. 2002 Sep;30(9):2022-9. doi: 10.1097/00003246-200209000-00011. PMID 12352035
- [Result] Cruzat V, Macedo Rogero M, Noel Keane K, Curi R, Newsholme P. Glutamine: Metabolism and Immune Function, Supplementation and Clinical Translation. Nutrients. 2018 Oct 23;10(11):1564. doi: 10.3390/nu10111564. PMID 30360490